CLINICAL TRIAL: NCT04108117
Title: Surgical and Oncologic Outcomes After Robotic Nipple Sparing Mastectomy and Immediate Reconstruction : an International Multicenter Pooled Analysis
Brief Title: Surgical and Oncologic Outcomes After Robotic Nipple Sparing Mastectomy and Immediate Reconstruction
Acronym: SORI
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Collaborators: European Institute of Oncology (Other); Changhua Christian Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyung Seok Park, MD, PhD, Clinical Associate Professor, Severance Hospital
Other Study IDs: 4-2019-0834
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Complications; Recurrence; Breast Neoplasms; Breast Cancer; BRCA1 Mutation; BRCA2 Mutation; Surgery; Surgery--Complications
Keywords: Robotic mastectomy; Breast neoplasms; Postoperative complications; Recurrence; Prognosis; Survivals; Nipple sparing mastectomy; Immediate reconstruction
MeSH Terms: conditions — Postoperative Complications; Recurrence; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic nipple sparing mastectomy group/RNSM: Cases or Patients who underwent robotic nipple-sparing mastectomy and immediate reconstruction are enrolled in this arm. Robotic nipple-sparing mastectomy should be performed using robotic surgical systems. Robotic surgical systems include da Vinci S,Si, X, Xi, and SP systems. Axillary or lateral incisions are used for this procedure. Immediate reconstruction includes tissue expander insertion, direct-to-implant, latissimus dorsi flap, transverse abdominis rectus muscle flap, or deep inferior epigastric perforators flap. Cases with robotic mastectomy without immediate reconstruction are excluded.
  The estimated sample size for this arm is 300 cases.
  Interventions: Procedure: Robotic nipple sparing mastectomy
- Conventional nipple sparing mastectomy group/CNSM: Cases or Patients who underwent conventional nipple-sparing mastectomy and immediate reconstruction are enrolled in this arm. Conventional nipple-sparing mastectomy should not be performed using robotic or endoscopic surgical systems. Axillary or lateral incisions that are similar to incisions in robotic nipple-sparing mastectomy are not allowed. Other than axillary or lateral incisions can be performed for this procedure. Immediate reconstruction includes tissue expander insertion, direct-to-implant, latissimus dorsi flap, transverse abdominis rectus muscle flap, or deep inferior epigastric perforators flap. Cases with nipple-sparing mastectomy without immediate reconstruction are excluded.
  The estimated sample size for this arm is 300 cases.

INTERVENTIONS:
Procedure: Robotic nipple sparing mastectomy — Robotic nipple sparing mastectomy means nipple sparing mastectomy performed using robotic surgical systems.
  Other Names: Robot-assisted nipple sparing mastectomy; Robot mastectomy; Robotic mastectomy; Hybrid robotic nipple sparing mastectomy; Robot-assisted nipple areolar complex and skin sparing mastectomy
  Groups: Robotic nipple sparing mastectomy group/RNSM

SUMMARY:
Robotic mastectomy with immediate reconstruction was introduced by Toesca et al. in 2015. Since then, several studies have reported the safety and feasibility of robotic nipple-sparing mastectomy with immediate reconstruction. However, most studies were conducted by single centers and had small samples. Furthermore, there is a lack of studies comparing surgical and oncologic outcomes between robotic nipple-sparing mastectomy and conventional nipple-sparing mastectomy. For this reason, this study evaluates surgical and oncologic outcomes of robotic nipple-sparing mastectomy with immediate reconstruction using international multi-center data.

DETAILED DESCRIPTION:
This study is an international multi-center pooled analysis using prospective and retrospective studies to evaluate surgical and oncologic outcomes of robotic nipple-sparing mastectomy with immediate reconstruction.

Raw data for robotic or conventional nipple-sparing mastectomy from Severance Hospital, Samsung Medical Center, the European Institute of Oncology, Changhua Christian Hospital, and Gustave Roussy is collected. Among them, Severance Hospital takes the lead at performing analysis from the data. Storage and disposal of patients' records are managed by each researcher. In the analysis process, although the collaborators can request records from Severance Hospital if necessary, they are only supposed to be provided computerized data which were originally clinical data from patients who already ended treatments. In this case, individual identifying data and medical records are not shown.

Clinicopathologic variables including operation times, hospital stay, medical history, smoking history, family history, BMI, menopausal status, specimen weight, TNM stage, grade, histological type, estrogen receptor, progesterone receptor, HER2, Ki 67, and perivascular involvement are analyzed.

Postoperative complications within 30 days are collected and classified by the Clavien-Dindo grade. Locoregional recurrence-free survival and local and systemic recurrences are examined. Patients whose data have been retrospective for at least one month are to be examined.

Patient's and surgeon's satisfaction using Breast Q is evaluated. Categorical variables are examined using the chi-square test or Fisher's exact test if indicated.

Continuous variables are examined using the independent t-test or ANOVA if indicated.

The estimated sample size from the four institutions is about 300 cases for robotic nipple-sparing mastectomy and matched cases for conventional nipple-sparing mastectomy.

Propensity matching analysis is applied to reduce confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent nipple sparing mastectomy and immediate reconstruction
* Women with early breast cancer
* Women with germline BRCA 1/2 mutation or germline mutations in genetic susceptibility genes
* Women with interstitial mastopathy
* Women with risk-reducing mastectomy or contralateral mastectomy

Exclusion Criteria:

* Male patients
* Women with stage IV disease at diagnosis
* Women who underwent previous breast cancer surgery
* Women who received prior radiotherapy for the ipsilateral breast

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent nipple-sparing mastectomy between 2016 and 2020 at Severance Hospital, Seoul, Korea.
  Patients who underwent nipple-sparing mastectomy between 2016 and 2020 at Samsung Medical Center, Seoul, Korea.
  Patients who underwent nipple sparing mastectomy between 2014 and 2019 at European Institute of Oncology, Milan, Italy.
  Patients who underwent nipple-sparing mastectomy between 2017 and 2019 at Changhua Christian Hospital, Changhua City, Taiwan.
  Patients who underwent nipple-sparing mastectomy between 2015 and 2019 at Gustave Roussy, Paris, France.
Sampling Method: Non-Probability Sample
Enrollment: 659 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Postoperative complication rates in 30 days | Postoperative 30 days
  Postoperative complication rates are calculated as total number of postoperative complication cases per total operation cases.
Clavien-Dindo grade of postoperative complications | Postoperative 30 days
  Clavien-Dindo grade of postoperative complications is evaluated. The highest grade of postoperative complications are used for the analysis.
Nipple necrosis rates | Postoperative 30 days
  Nipple necrosis rates are calculated as number of total nipple necrosis cases per total operation cases.
Recurrence free survival (RFS) | Postoperative 5 years
  Events of RFS includes locoregional recurrence, distant recurrence, and death. Contralateral breast cancer and second primary malignancy are considered to be censored data.

SECONDARY OUTCOMES:
Operation times | Time during operation
  Mastectomy time or reconstruction time
Locoregional recurrence-free survival (LRFS) | Postoperative 5 years
  In breast tumor recurrences (IBTR), regional recurrences including axillary, internal mammary, or supraclavicular lymph node recurrences, and death without any cause are events of locoregional recurrence-free survival. Five year LRFS is measured. Distant metastasis, contralateral breast cancer and second primary malignancy are considered to be censored data.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Seok Park, MD, PhD, Principal Investigator — Severance Hospital; Antonio Toesca, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
After completion of this study, IPD can be considered based on the decision of the study steering comittee.

REFERENCES:
- [Background] Toesca A, Peradze N, Manconi A, Galimberti V, Intra M, Colleoni M, Bonanni B, Curigliano G, Rietjens M, Viale G, Sacchini V, Veronesi P. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast. 2017 Feb;31:51-56. doi: 10.1016/j.breast.2016.10.009. Epub 2016 Nov 2. PMID 27810700
- [Background] Park HS, Kim JH, Lee DW, Song SY, Park S, Kim SI, Ryu DH, Cho YU. Gasless Robot-Assisted Nipple-Sparing Mastectomy: A Case Report. J Breast Cancer. 2018 Sep;21(3):334-338. doi: 10.4048/jbc.2018.21.e45. Epub 2018 Sep 20. PMID 30275863
- [Background] Galimberti V, Morigi C, Bagnardi V, Corso G, Vicini E, Fontana SKR, Naninato P, Ratini S, Magnoni F, Toesca A, Kouloura A, Rietjens M, De Lorenzi F, Vingiani A, Veronesi P. Oncological Outcomes of Nipple-Sparing Mastectomy: A Single-Center Experience of 1989 Patients. Ann Surg Oncol. 2018 Dec;25(13):3849-3857. doi: 10.1245/s10434-018-6759-0. Epub 2018 Sep 17. PMID 30225833
- [Background] Toesca A, Peradze N, Galimberti V, Manconi A, Intra M, Gentilini O, Sances D, Negri D, Veronesi G, Rietjens M, Zurrida S, Luini A, Veronesi U, Veronesi P. Robotic Nipple-sparing Mastectomy and Immediate Breast Reconstruction With Implant: First Report of Surgical Technique. Ann Surg. 2017 Aug;266(2):e28-e30. doi: 10.1097/SLA.0000000000001397. No abstract available. PMID 28692558
- [Background] Toesca A, Peradze N, Manconi A, Nevola Teixeira LF. Reply to the letter to the editor "Robotic-assisted Nipple Sparing Mastectomy: A feasibility study on cadaveric models" by Sarfati B. et al. J Plast Reconstr Aesthet Surg. 2017 Apr;70(4):558-560. doi: 10.1016/j.bjps.2016.12.022. Epub 2017 Jan 23. No abstract available. PMID 28153430
- [Background] Lai HW, Wang CC, Lai YC, Chen CJ, Lin SL, Chen ST, Lin YJ, Chen DR, Kuo SJ. The learning curve of robotic nipple sparing mastectomy for breast cancer: An analysis of consecutive 39 procedures with cumulative sum plot. Eur J Surg Oncol. 2019 Feb;45(2):125-133. doi: 10.1016/j.ejso.2018.09.021. Epub 2018 Oct 17. PMID 30360987
- [Background] Lai HW, Lin SL, Chen ST, Chen SL, Lin YL, Chen DR, Kuo SJ. Robotic Nipple-sparing Mastectomy and Immediate Breast Reconstruction with Gel Implant. Plast Reconstr Surg Glob Open. 2018 Jun 11;6(6):e1828. doi: 10.1097/GOX.0000000000001828. eCollection 2018 Jun. PMID 30276055
- [Background] Lai HW. Robotic Nipple-Sparing Mastectomy and Immediate Breast Reconstruction with Gel Implant. Ann Surg Oncol. 2019 Jan;26(1):53-54. doi: 10.1245/s10434-018-6711-3. Epub 2018 Aug 25. No abstract available. PMID 30145648
- [Background] Lai HW, Lin SL, Chen ST, Lin YL, Chen DR, Pai SS, Kuo SJ. Robotic nipple sparing mastectomy and immediate breast reconstruction with robotic latissimus dorsi flap harvest - Technique and preliminary results. J Plast Reconstr Aesthet Surg. 2018 Oct;71(10):e59-e61. doi: 10.1016/j.bjps.2018.07.006. Epub 2018 Aug 2. No abstract available. PMID 30122600
- [Background] Lai HW, Chen ST, Lin SL, Chen CJ, Lin YL, Pai SH, Chen DR, Kuo SJ. Robotic Nipple-Sparing Mastectomy and Immediate Breast Reconstruction with Gel Implant: Technique, Preliminary Results and Patient-Reported Cosmetic Outcome. Ann Surg Oncol. 2019 Jan;26(1):42-52. doi: 10.1245/s10434-018-6704-2. Epub 2018 Aug 14. PMID 30109537
- [Background] Lai HW, Chen ST, Lin SL, Lin YL, Wu HK, Pai SH, Chen DR, Kuo SJ. Technique for single axillary incision robotic assisted quadrantectomy and immediate partial breast reconstruction with robotic latissimus dorsi flap harvest for breast cancer: A case report. Medicine (Baltimore). 2018 Jul;97(27):e11373. doi: 10.1097/MD.0000000000011373. PMID 29979425
- [Background] Sarfati B, Struk S, Leymarie N, Honart JF, Alkhashnam H, Tran de Fremicourt K, Conversano A, Rimareix F, Simon M, Michiels S, Kolb F. Robotic Prophylactic Nipple-Sparing Mastectomy with Immediate Prosthetic Breast Reconstruction: A Prospective Study. Ann Surg Oncol. 2018 Sep;25(9):2579-2586. doi: 10.1245/s10434-018-6555-x. Epub 2018 Jun 29. PMID 29959612
- [Background] Sarfati B, Struk S, Leymarie N, Honart JF, Alkhashnam H, Kolb F, Rimareix F. Robotic Nipple-Sparing Mastectomy with Immediate Prosthetic Breast Reconstruction: Surgical Technique. Plast Reconstr Surg. 2018 Sep;142(3):624-627. doi: 10.1097/PRS.0000000000004703. PMID 29879007
- [Background] Sarfati B, Honart JF, Leymarie N, Rimareix F, Al Khashnam H, Kolb F. Robotic da Vinci Xi-assisted nipple-sparing mastectomy: First clinical report. Breast J. 2018 May;24(3):373-376. doi: 10.1111/tbj.12937. Epub 2017 Dec 18. PMID 29251382
- [Background] Sarfati B, Honart JF, Leymarie N, Kolb F, Rimareix F. Robotic-assisted Nipple Sparing Mastectomy: A feasibility study on cadaveric models. J Plast Reconstr Aesthet Surg. 2016 Nov;69(11):1571-1572. doi: 10.1016/j.bjps.2016.08.007. Epub 2016 Sep 8. No abstract available. PMID 27665275
- [Result] Park HS, Lee J, Lai HW, Park JM, Ryu JM, Lee JE, Kim JY, Marrazzo E, De Scalzi AM, Corso G, Montemurro F, Gazzetta G, Pozzi G, Toesca A. Surgical and Oncologic Outcomes of Robotic and Conventional Nipple-Sparing Mastectomy with Immediate Reconstruction: International Multicenter Pooled Data Analysis. Ann Surg Oncol. 2022 Oct;29(11):6646-6657. doi: 10.1245/s10434-022-11865-x. Epub 2022 May 18. PMID 35583693